CLINICAL TRIAL: NCT01123135
Title: The Effect of Vaginal Estrogen Cream on Subjective and Objective Symptoms of Urodynamic Stress Incontinence
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to determine a suitable placebo.
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-6434
Record Dates: First submitted 2010-05-06; First posted 2010-05-14 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Stress Urinary Incontinence
Keywords: urodynamic stress incontinence; postmenopausal women
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal ERT (Active Comparator): Vaginal ERT cream 1 gm at bed time 3 times a week
  Interventions: Drug: Vaginal ERT
- Placebo (Placebo Comparator): 1gm of placebo at bed time 3 times a week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vaginal ERT — 1gm of estrogen vaginal cream [EVC] at bed time 3 times a week
  Arms: Vaginal ERT
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double blinded placebo controlled trial over a period of 3 months. Study subjects will be randomized into 2 groups: Those receiving drug (1gm of estrogen vaginal cream [EVC] at bed time 3 times a week), and those receiving placebo.

DETAILED DESCRIPTION:
1. This will be a randomized, double blinded placebo controlled trial over a period of 3 months. Study subjects will be randomized into 2 groups: Those receiving drug (1gm of estrogen vaginal cream [EVC] at bed time 3 times a week), and those receiving placebo. Study subjects will be patients diagnosed with stress urinary incontinence by urodynamic evaluation. They will have filled out the IIQ-7 and UDI-6 validated questionnaires as is routine for all patients being evaluated for stress incontinence. After enrollment and informed consent, their initial screening will include a Pap smear for vaginal maturation.
2. Subjects will then be seen at 4, 8 and 12 weeks. At each visit, they will turn in their medication tubes and receive new study medication. They will also be screened for any adverse reaction to the study medication at each visit.
3. At the end of the study period, the subjects will fill out the same validated questionnaire as they did at the beginning of the study and they will also have their urethral pressure profile and PAP smear repeated.
4. The urethral pressure profile is part of the standard complex urodynamic testing that all patients undergo for evaluation and diagnosis of urodynamic stress incontinence. Urethral Pressure Profile is a technique used to provide information about the ability of the urethra to prevent leakage. The Urethral Pressure Profile is a specific study, in which a special design catheter is pulled through the urethra at a slow, continuous rate. The resulting "bell shaped" curve illustrates the function of the urethra from the beginning of the bladder neck out through the meatus.
5. The placebo cream will be a pharmacologically inert formulation which will be packaged similarly to the active premarin cream and visually indistinguishable from the active drug to both the study subjects and researchers.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Postmenopausal women (No menses for a minimum period of 1 year)
* Urodynamic stress urinary incontinence

Exclusion Criteria:

* History of breast or uterine cancer
* History of venous thrombolic event
* Hormone replacement therapy within 3 months of study
* Sensitivity or allergy to premarin cream
* Current use of any medications for urge or stress incontinence
* Prior surgery for stress incontinence
* Overactive bladder or Detrussor instability
* Active vaginal/ bladder infection (patients will be treated and have a negative test for cure in order to be enrolled in the study)
* History of pelvic or vaginal radiation therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the effects of vaginal estrogen replacement versus placebo on the subjective improvement of stress urinary incontinence symptoms with the use of validated questionnaires. | Exam at baseline and 12 weeks

SECONDARY OUTCOMES:
Determine effects of vaginal ERT vs placebo on objective improvement in urethral function by comparing pre and post treatment urethral closure pressures. Determine incidence of UTIs at the beginning of study compared to the end of the study. | Exam at baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Principal Investigator — UCI Medical Center
Locations (1):
- UC Irvine Women's Healthcare, Orange, California, United States